CLINICAL TRIAL: NCT00694200
Title: Vinorelbine Metronomic Plus Bevacizumab as Salvage Therapy for Patients With Metastatic Breast Cancer. A Multicenter Phase II Study
Brief Title: Vinorelbine Metronomic Plus Bevacizumab as Salvage Therapy for Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not reached the statistical hypothesis at the interim analysis
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/08.03
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; chemotherapy; anti-angiogenesis therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Vinorelbine metronomic + bevacizumab
  Interventions: Drug: Vinorelbine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine per os 50 mg 3 times a week
  Other Names: Navelbine
Drug: Bevacizumab — Bevacizumab 10 mg/kg IV every 14 days
  Other Names: Avastin

SUMMARY:
To evaluate the efficacy of metronomic oral vinorelbine taken three times a week without break plus bevacizumab as salvage treatment in patients with metastatic breast cancer.

DETAILED DESCRIPTION:
Continuous administration of oral vinorelbine, given three times a week (metronomic) is feasible and exceptionally well tolerated at doses up to 50 mg. Early results show activity against refractory tumors and provide evidence towards clinical proof of efficacy for metronomic chemotherapy. Recently, initial therapy of metastatic breast cancer with paclitaxel plus bevacizumab demonstrated prolonged progression-free survival, as compared with paclitaxel alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed metastatic breast adenocarcinoma
* At least one previous chemotherapy regimen for metastatic breast cancer
* Age 18-75 years
* Measurable disease as defined by the presence of at least one measurable lesion (except bone metastases, ascites or pleural effusions)
* Performance status (WHO) 0-2
* Adequate liver function(serum bilirubin <1.5 times the upper normal limit, AST and ALT <2.5 times the upper normal limit in the absence of demonstrable liver metastases, or <5 times the upper normal limit in the presence of liver metastases), adequate renal function (serum creatinine <1.5 times the upper normal limit) and bone marrow (neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L) function
* No radiation of measurable disease (except brain metastases)
* No progressive brain metastases according to clinical or radiological criteria
* No brain metastases without prior radiation therapy
* Written informed consent

Exclusion Criteria:

* Patient unable to take oral medication
* Active infection
* History of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* History of stroke
* Anticoagulation therapy (except of low dose aspirin <325mg)
* Other invasive malignancy except nonmelanoma skin cancer
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Response rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Duration of response | 1 year
Progression free survival | 1 year
Overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (9):
- Greece (9):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki